CLINICAL TRIAL: NCT06506981
Title: Association Between Electrolyte Intake and Growth Trajectories in Premature Newborns : a Retrospective Population-based Study Between January 2023 and December 2023 at the Regional Maternity Hospital of Nancy
Brief Title: Impact of Electrolyte Intake (Sodium, Phosphorus) on the Growth of Premature Newborns
Acronym: ELECTROGRO
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Jean-Michel HASCOET, Pofessor, Central Hospital, Nancy, France
Other Study IDs: 2024PI124
Record Dates: First submitted 2024-07-10; First posted 2024-07-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Postnatal Growth Disorder
Keywords: parenteral nutrition; enteral nutrition; electrolyte intake; premature newborn; growth trajectory
MeSH Terms: conditions — Hyperphagia; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Extrauterine growth restriction (EUGR) is a common complication in the medical management of premature newborns. The long-term consequences of EUGR are weight and height restriction, metabolic disorders, and neurodevelopmental disorders. The main risk factor for EUGR is nutritional deficiency, particularly protein and energy. Additionally, appropriate intakes of electrolytes, particularly sodium and phosphorus, are essential to promote harmonious growth. Adequate sodium intake is essential to ensure satisfactory growth, especially in premature babies due to their higher body water content. Adequate phosphorus intake is also essential because of its involvement in the formation of lean mass, with sufficient protein intake, and in phosphocalcic metabolism.

At the Regional University Maternity of Nancy, parenteral and enteral nutrition prescriptions for each premature newborn are made using the Logipren® prescription assistance software, based on ESPGHAN recommendations. Despite this theoretical security, it seems that they are not strictly respected. At the same time, premature newborns typically show weight loss often greater than -1 z-score.

The objective of this research is to study the impact of electrolyte intake (sodium and phosphorus) on growth trajectories and the incidence of EUGR in premature newborns discharged from the Nancy Maternity Hospital in 2023. The secondary criteria are to describe sodium, phosphorus, protein and calorie intake and compliance with ESPGHAN recommendations; assess the true prevalence of stunting in our study population; and the impact of meeting electrolyte intake recommendations on children's growth trajectory, taking into account protein and calorie intake.

ELIGIBILITY:
Inclusion Criteria:

* Neonates born between January 1st 2023 and December 31st 2023
* Neonates born before 37 SA
* Neonates hospitalized at the Nancy Maternity Hospital in Neonatology

Exclusion Criteria:

* Neonates transferred at the Nancy Maternity Hospital after 48 first hours of life

Ages: 1 Day to 30 Days | Sex: All
Age Groups: Child
Study Population: All premature neonates born between January 1st 2023 and December 31st 2023 who were hospitalized at the Nancy Maternity Hospital in Neonatology
Sampling Method: Non-Probability Sample
Enrollment: 684 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Relationship between electrolyte intake (sodium and phosphorus) and the occurrence of Growth retardation (EUGR) in preterm neonates | 30 days
  Sodium and phosphorus intake according to the recommendations of the European Society of Pediatric Gastroenterology, Hepatology and Nutrition (ESPGHAN) for parenteral nutrition. The hypothesis is that electrolyte intakes lower than the ESPGHAN recommendation should induce an EUGR defined as a loss of one standard deviation according to the reference growth curves (Fenton reference).

SECONDARY OUTCOMES:
Sodium intake descriptive study | 30 days
  Total daily sodium intake, in mmol/Kg/d, during the first 30 days, or up to the date of discharge if before 30 days, according to ESPGHAN recommendations for parenteral nutrition.
Phosphorus intake descriptive study | 30 days
  Total daily phosphorus intake, in mmol/Kg/d, during the first 30 days, or up to the date of discharge if before 30 days, according to ESPGHAN recommendations for parenteral nutrition.
Protein intake descriptive study | 30 days
  Total daily protein intake, in g/Kg/d, during the first 30 days, or up to the date of discharge if before 30 days, according to ESPGHAN recommendations for parenteral nutrition.
Calories intake descriptive study | 30 days
  Total daily calories intake, in kCal/Kg/d, during the first 30 days, or up to the date of discharge if before 30 days, according to ESPGHAN recommendations for parenteral nutrition.
Weight growth descriptive study | 30 days
  Daily weight trajectory in grams/Kg/d during the first 30 days or up to the date of discharge if before 30 days.
Weight growth according to reference curve for the population | 30 days
  Weight trajectory according to Fenton reference curves in z-score
Relationship between sodium intake and the occurrence of EUGR in preterm neonates after adjusting on protein and calorie intake | 30 days
  Correlation between eletrolyte intake and growth trajectory
Relationship between phosphorus intake and the occurrence of EUGR in preterm neonates after adjusting on protein and calorie intake | 30 days
  Correlation between eletrolyte intake and growth trajectory

CONTACTS AND LOCATIONS:
Locations (1):
- Maternity Hospital CHRU, Nancy, Lorraine, France